CLINICAL TRIAL: NCT02220140
Title: Resilience for Young People With Attention Deficit Hyperactivity Disorder (ADHD) - a Randomized Controlled Trial of a Brief Intervention Program.
Brief Title: Resilience for Young People With ADHD - a Randomized Controlled Trial of a Brief Intervention Program.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DK-res-adhd
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Service as usual
- Intervention group (Experimental): Participants are offered access to the web based resilience program and are invited to join a short introduction course.
  Interventions: Behavioral: The Resilience Program

INTERVENTIONS:
Behavioral: The Resilience Program — See the CONSORT trial protocol at http://myresilience.org/ at the subsite 'about us'.
  Arms: Intervention group

SUMMARY:
In this project we invite 8.000 young persons (age 18-27) in Denmark and to participate in a randomized controlled intervention study where we aim to test the effectiveness of a web based knowledge and inspiration program about resilience for children, adolescents and adults (called myresilience.org). The complete CONSORT trial protocol is available at http://myresilience.org/ at the subsite 'about us'.

DETAILED DESCRIPTION:
The complete CONSORT trial protocol is available at http://myresilience.org/ at the subsite 'about us'.

ELIGIBILITY:
Inclusion Criteria:

A random sample with 8.000 patients registered in the Danish National Patient Register:

* Age 18-27
* ADHD diagnosis

Exclusion Criteria:

• Request for legal protection against contacts from researchers.

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8000 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Adult ADHD Self-Report Scale (ASRS-v1.1) | Follow-up will be on the average 1 year after intervention
  The Symptom Checklist is an instrument consisting of the eighteen Diagnostic and Statistical Manual criteria (DSM-IV). Six of the eighteen questions were found to be the most predictive of symptoms consistent with ADHD. These six questions are the basis for the ASRS v1.1. The measure is a number score.
  The ASRS-v1.1 will be administered to all participants before and 1 year after the intervention.

SECONDARY OUTCOMES:
The 12-item General Health Questionnaire (GHQ-12) | Follow-up will be on the average 1 year after intervention
  The GHQ-12 is a widely used standard Health Questionnaire. The GHQ-12 will be administered to all participants before and 1 year after the intervention.
  The measure is a number score.

OTHER OUTCOMES:
Youth education attrition | December 2016

CONTACTS AND LOCATIONS:
Overall Officials: Poul L Bak, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

REFERENCES:
- See also: See the CONSORT trial protocol at the subsite 'about us' — http://myresilience.org/